CLINICAL TRIAL: NCT02183779
Title: Rôle Des Acides Epoxy-eicosatriénoïques et du Monoxyde d'Azote Dans l'hyperhémie Post-occlusive cutanée Digitale et la réponse cutanée au Froid Dans le phénomène de Raynaud Primaire
Brief Title: PORH and Response to Cold in Raynaud's Phenomenon.
Acronym: REFRAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DCIC 14 02
Record Dates: First submitted 2014-07-01; First posted 2014-07-08 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Raynaud Disease; Hyperemia; Cold
Keywords: post-occlusive hyperaemia; laser-speckle contrast imaging; epoxyeicosatrienoic acid; nitrous oxide
MeSH Terms: conditions — Raynaud Disease; Hyperemia; Common Cold | interventions — omega-N-Methylarginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reynaud (Experimental): patients with reynaud phenomena
  Interventions: Procedure: post-occlusive hyperemia; Procedure: cooling box; Drug: L-NMMA and Fluconazole dermic injection
- Healthy (Experimental): Healthy volunteers
  Interventions: Procedure: post-occlusive hyperemia; Procedure: cooling box; Drug: L-NMMA and Fluconazole dermic injection

INTERVENTIONS:
Procedure: post-occlusive hyperemia
Procedure: cooling box
Drug: L-NMMA and Fluconazole dermic injection

SUMMARY:
The main objective of the study is to determine if implication of epoxy-eicosatriénoïc acids (EETs) and NO during cutaneous post-occlusive hyperemia differs between patients with Raynaud phenomena and healthy volunteers, by studying hyperaemic postocclusive response after microinjection of fluconazole and L-NMMA at the dorsal side of the fingers.

DETAILED DESCRIPTION:
The main objective of the study is to determine if implication of epoxy-eicosatriénoïques acids (EETs) and NO during cutaneous post-occlusive hyperemia differs between patients with Raynaud phenomena and healthy volunteers, by studying hyperaemic postocclusive response after microinjection of fluconazole and L-NMMA at the dorsal side of the fingers.

Healthy controls and patients will undergo 3 visits

ELIGIBILITY:
Inclusion Criteria:

* Neither raynaud's phenomenon or chronic disease for healthy volunteers
* Raynaud's phenomenon without connective tissue disease for patients in the group "Raynaud"

Exclusion Criteria:

* History of axillary dissection , trauma or surgery
* History of thromboembolic disease or thrombophilia
* Minor or law-protected major
* Exclusion period in another study
* No affiliation to medicare
* Pregnant, parturient or breasting woman
* Concomitant serious disease: progressive cancer, liver failure, history of myocardial infarction less than 5 years, angor
* Smoking in the 6 last months
* Person deprived of liberty by a legal or administrative decision, person under legal protection
* Maximal annual indemnification reached.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-10 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
post occlusive hyperemia amplitude | day 1
  post-occlusive hyperemia amplitude (maximal amplitude in % of maximal vasodilatation and AUC) in sites NaCl, fluconazole and L-NMMA (intradermal microinjection)

SECONDARY OUTCOMES:
post occlusive hyperemia amplitude with anesthetic treatment | day1
  post-occlusive hyperemia amplitude (maximal amplitude in % of maximal vasodilatation and AUC) in sites NaCl, fluconazole and L-NMMA (intradermal microinjection) treated with anesthetic
cold-induced vasoconstriction amplitude | day 2
  cold-induced vasoconstriction amplitude (maximal amplitude in % of basal and AUC) in sites NaCl, fluconazole and L-NMMA (intradermal microinjection)
cold-induced vasoconstriction amplitude with anesthetic treatment | day 2
  cold-induced vasoconstriction amplitude (maximal amplitude in % of basal and AUC) in sites NaCl, fluconazole and L-NMMA (intradermal microinjection) with anesthetic local treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc CRACOWSKI, MD-PhD, Principal Investigator — INSERM + University Hospital Grenoble
Locations (1):
- Centre d'investigation clinique CIC1406, Grenoble Cedex9, France